CLINICAL TRIAL: NCT00081978
Title: A Randomized, Controlled, Partially Blinded Phase IIb Dose-Finding Trial of TMC125 in HIV-1 Infected Subjects With Documented Genotypic Evidence of Resistance to Currently Available NNRTIs and With at Least Three Primary PI Mutations
Brief Title: TMC125-C223: TMC125 in HIV-1 Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CR006736
Record Dates: First submitted 2004-04-28; First posted 2004-04-30 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: HIV Infection
Keywords: HIV infection; TMC125; Non-nucleoside reverse transcriptase inhibitor, TMC125-C223
MeSH Terms: conditions — HIV Infections | interventions — etravirine

INTERVENTIONS:
Drug: TMC125

SUMMARY:
The purpose of this study is to investigate the ability of TMC125, a Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI), to lower the amount of virus in your blood when administered twice daily for 48 weeks.

DETAILED DESCRIPTION:
TMC125 will be given in addition to a combination of anti-HIV drugs that have been selected specifically for you by your doctor. There are three treatment groups in the study. One group will be given a dosage of TMC125, 400 mg twice daily. Another will be given 800 mg twice daily. The third group, a control arm, will not receive TMC125 (formulation TF035). The safety, tolerability and pharmacokinetics (determinations of the concentration of drug in your blood and its evolution over time) of TMC125 will also be evaluated in this study. Patients who have known resistance to NNRTIs and 3 or more protease inhibitor (PI) mutations may be eligible to participate. One-hundred-fifty (150) patients will be enrolled into this study. TMC125, 400mg twice daily for 48 weeks; TMC125, 800mg twice daily for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 plasma viral load at screening >1000 copies/ml
* Documented genotypic evidence of resistance to currently available NNRTIs
* Previous NRTI experience for at least 3 months
* 3 primary PI mutations at screening

Exclusion Criteria:

* Chronic HBV and/or HCV with elevated liver function tests > 3x upper normal limits
* Any grade 3 or 4 toxicity according to the ACTG grading severity list (except for grade 3 glucose and asymptomatic triglyceride/cholesterol grade 3 or 4 elevation)
* Previous permanent discontinuation of any NNRTI due to cutaneous events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2004-03; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of the trial is to evaluate the dose-response relationship of antiviral activity at 24 weeks within the two TMC125 dose regimens.

SECONDARY OUTCOMES:
Evaluate the antiviral activity, safety and tolerability of TMC125, immunologic changes, changes in viral genotype and drug suseptibility, PK of TMC125 and compare antiviral effect among treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- [Result] Cohen CJ, Berger DS, Blick G, Grossman HA, Jayaweera DT, Shalit P, Thompson M, Peeters M, de Bethune MP, Voorspoels E, Mack R, Woodfall B. Efficacy and safety of etravirine (TMC125) in treatment-experienced HIV-1-infected patients: 48-week results of a phase IIb trial. AIDS. 2009 Jan 28;23(3):423-6. doi: 10.1097/QAD.0b013e32831c5040. PMID 19114852